CLINICAL TRIAL: NCT04279028
Title: Testing Different Modes of Cognitive Behavior Therapy
Acronym: CBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, James W Griffith, Associate Professor of Medical Social Sciences, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00210885
Record Dates: First submitted 2020-02-14; First posted 2020-02-20 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Depression; Literacy
MeSH Terms: conditions — Depression; Literacy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are told they will receive one of two forms of CBT. They will not receive details about the other group.
  The outcomes assessor will have no information about group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard CBT (Active Comparator): Standard CBT, 12 sessions each lasting 45 minutes
  Interventions: Behavioral: Standard CBT
- Adapted CBT (Experimental): Adapted CBT, 12 sessions each lasting 45 minutes
  Interventions: Behavioral: Adapted CBT

INTERVENTIONS:
Behavioral: Adapted CBT — ACBT is derived from traditional CBT principles, but eliminates the text-heavy requirements. Traditional CBT incorporates the use of complex worksheets and a lengthy workbook, whereas ACBT replaces these skill learning activities with simpler, straightforward exercises that are practiced in session along with the therapist. This "real world" practice eliminates the need for reading and writing as part of CBT while simultaneously recapitulating how the patient would actually implement CBT procedures. In session exercises will mirror that of standard CBT practices. For example, they could include lessons in goal setting, distinguishing situations, moods, and thoughts, and experiments to test underlying assumptions. Participants will be assigned paper-free homework assignments.
  Arms: Adapted CBT
Behavioral: Standard CBT — CBT involves the therapist and client working to identify and change negative beliefs and thoughts, replacing them with more accurate and balanced thoughts. CBT for Depression will be conducted according to standard manuals and incorporate the use of a common workbook used within CBT sessions. As per standard practice, participants will be assigned worksheets from their workbook used both in session and as homework assignments.
  Arms: Standard CBT

SUMMARY:
The purpose of this study is to test a novel behavioral treatment - Adapted Cognitive-Behavior Therapy (ACBT) - against standard Cognitive Behavior Therapy (CBT). The goal of the study is to determine if ACBT confers improved outcomes for women with depression and low literacy. Depression is a serious women's health issue. According to the World Health Organization, depression is the leading cause of disability worldwide with females reporting symptoms of depression at almost twice the rate of males. This study will provide pilot data to enable us to determine the effect size needed to detect a between-groups change in depression scores. The overall impact of this study will be empirical support for a novel form of treatment for women with depression, who also may lack adequate literacy, educational, or cognitive ability required to benefit from standard CBT.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. female
3. diagnosis of major depressive disorder (MDD) according to DSM-5 (Diagnostic and Statistical Manual-5) (and no specifiers that pertain to exclusionary criteria (e.g. MDD with psychotic features)
4. able and willing to give informed consent
5. able to communicate in English
6. willingness to be randomized to therapy
7. willing to complete all study assessments
8. at baseline, no plans to move from the Chicago area during the duration of the study

Exclusion Criteria:

1. history of bipolar disorder
2. history of psychosis
3. current substance use disorder of moderate or severe level of severity
4. suicidal intentions or actions within the past three months
5. known neurologic disease (e.g., multiple sclerosis, Parkinson's disease, cerebrovascular accident) and/or cognitive or neurologic impairment (e.g., Alzheimer's disease)
6. current participation in other psychotherapy (not including psychiatric appointments pertaining to medication management)
7. inadequate vision or hearing to interact with study materials
8. being a prisoner, detainee, or being in police custody
9. any current involvement in litigation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
PROMIS Depression: Post-treatment (defined as completing 12 therapy session) | Post-treatment which is within 2 weeks after final therapy session (i.e. estimated 12-14 weeks after initial intake interview)
  Defined remission of MDD (partial or full) established by PROMIS (Patient-Reported Outcomes Measurement Information System).
PROMIS Depression: : 3-month follow-up (defined as 3 months after the last (i.e., 12th) session of cognitive behavior therapy. | 3-month follow up (i.e., 3 months after the end of treatment)
  Defined remission of MDD (partial or full) established by PROMIS.

SECONDARY OUTCOMES:
World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0): Post-treatment (defined as completing 12 sessions of therapy; this will occur an estimated 12-14 weeks after initial intake interview) | Post-treatment which is within 2 weeks after final therapy session (i.e. estimated 12-14 weeks after initial intake interview)
  The 12-item WHODAS 2.0 is a measure of functional impairment. Higher scores indicate a higher level of impairment.
  The scores for each item range from 0-4; the WHO scoring algorithm converts the summed score to a 0-100% score.
  The post-treatment score will be compared to baseline to quantify reduction of impairment after treatment.
World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0): 3-month follow-up (defined as 3 months after the end of treatment) | 3-month follow up (i.e., 3 months after the end of treatment)
  The 12-item WHODAS 2.0 is a measure of functional impairment. Higher scores indicate a higher level of impairment.
  The scores for each item range from 0-4; the WHO scoring algorithm converts the summed score to a 0-100% score.
  The 3-month follow-up score will be compared to baseline to quantify reduction of impairment after treatment.

OTHER OUTCOMES:
Patient Global Impression of Change (PGIC): Post-treatment (defined as completing 12 sessions of therapy; this will occur an estimated 12-14 weeks after initial intake interview) | Post-treatment which is within 2 weeks after final therapy session (i.e. estimated 12-14 weeks after initial intake interview)
  Allows for the participant to indicate change in either direction (ie, much better, much worse)
Patient Global Impression of Change (PGIC) 3-month follow-up (defined as 3 months after the end of treatment) | 3-month follow up (i.e., 3 months after the end of treatment)
  Allows for the participant to indicate change in either direction (ie, much better, much worse)
California Psychotherapy Alliance Scale - Participant version short-form - Post-treatment (defined as completing 12 sessions of therapy; this will occur an estimated 12-14 weeks after initial intake interview) | Post-treatment which is within 2 weeks after final therapy session (i.e. estimated 12-14 weeks after initial intake interview)
  Measures four independent dimensions of the therapeutic relationship

CONTACTS AND LOCATIONS:
Locations (1):
- James W. Griffith, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No